CLINICAL TRIAL: NCT06346275
Title: Effect of Acupuncture on the Gait Disturbance and Hemodynamic Changes in the Prefrontal Cortex: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of Acupuncture on the Gait Disturbance and Hemodynamic Changes in the Prefrontal Cortex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Zhenmei Hong, Principal Investigator, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3rdZhejiangCMU-11
Record Dates: First submitted 2024-03-24; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Cognitive rehabilitation therapy: The cognitive training system (JZ-RZ-1020, Extreme Medical Technology, Hangzhou, China) will be used to help develop personalized rehabilitation plans for one-on-one training based on the cognitive function of each patient. The trainings include memory, hand eye reinforcement, attention, reaction. Patients are treated for 30 minutes each time and 5 times a week for 8 weeks.
  Interventions: Procedure: Acupuncture
- Acupuncture group (Experimental): Acupoints: Baihui (GV20), Sishencong (EX-HN1), Fengchi (GB20), Taixi (KI3), Zusanli (ST36), Sanyinjiao (SP6), Neiguan (PC6), and Shenmen (HT7).
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupoints: Baihui (GV20), Sishencong (EX-HN1), Fengchi (GB20), Taixi (KI3), Zusanli (ST36), Sanyinjiao (SP6), Neiguan (PC6), and Shenmen (HT7).

SUMMARY:
Background: Alzheimer's disease (AD) is characterized by cognitive impairment and behavioral impairment, and increasing attention is paid in the gait of AD patients. The aim of this randomized controlled trial (RCT) is to explore the effect of acupuncture on the cognitive function, gait performance, and hemodynamic changes in the prefrontal cortices.

Methods: In this RCT, a total of 108 AD patients will be randomly assigned into acupuncture group or control group for 8 weeks. The primary outcome will be Three-dimensional gait analysis and cerebral hemodynamics using functional near-infrared spectroscopy (fNIRS). Secondary outcomes include Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), and Barthel Index (BI).

Discussion: This trial is expected to explore the effect of acupuncture on cognitive function, gait performance, and hemodynamic changes in the prefrontal cortices for AD patients.

DETAILED DESCRIPTION:
This study aims to assess the clinical effect of acupuncture on gait performance in AD patients and to examine the acupuncture effect on cerebral cortices by identifying hemodynamic changes that occur in the prefrontal cortices using the fNIRS technique.

ELIGIBILITY:
The inclusion criteria are as follows:

1. Aged 40-85 years old;
2. Meeting the mentioned-above diagnostic criteria from traditional Chinese medicine and Western medicine;
3. With mild to moderate dementia (CDR=0.5, 1.0, or 2.0 points);
4. Hachinski Ischemic Scale (HIS) ≤ 4 points;
5. Hamilton Depression Rating Scale (HAMD) < 20 points;
6. Without severe bone and joint diseases and able to walk independently;
7. Able to conduct vision and hearing tests;
8. Volunteering to participate in this trial and signing an informed consent form. Exclusion criteria

The exclusion criteria are as follows:

1. Dementia caused by other systemic or neurological diseases, such as central nervous system infections, post-traumatic dementia, Parkinson's disease dementia;
2. Suffering from acute illness, upper limb extrapyramidal stiffness, neurological or psychiatric disorders (except cognitive impairment);
3. With medical history that interferes with cognitive function assessment, such as past history of psychiatric drug abuse, drug addiction within the past 5 years, and alcohol abuse;
4. Afraid of acupuncture and cannot accept acupuncture treatment;
5. Currently participating in other clinical trial that affects the outcome evaluation of this trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional gait analysis | Assessments will be performed before the treatments, at 4 weeks after treatments, and at 8 weeks after treatments.
  Vicon's Nexus system detects gait parameters and kinematic parameters, including step length, stride, pace, step width, step frequency, single/double stand phase, turning (time and number of steps required for turning), swing phase.
Cerebral hemodynamics | Assessments will be performed before the treatments, at 4 weeks after treatments, and at 8 weeks after treatments.
  A total of 22 channels are configured using 8 emitters and 8 detectors, with each light source emitting three wavelengths (780 nm, 805 nm, and 830 nm) of light, and the original intensity signal is recorded at a sampling frequency of 13.33Hz. Patients need to try to keep the head fixed during the walking.

SECONDARY OUTCOMES:
Mini-Mental State Examination | Assessments will be performed before the treatments, at 4 weeks after treatments, and at 8 weeks after treatments.
  MMSE is a 30-point questionnaire, and 1 point is assigned for each correct answer. Testing scores are closely related to education level, and the standard for dividing the normal threshold is >17 points for patients with illiteracy, >20 points for patients with primary school, >22 points for patients with secondary school, and >23 points for patients with junior college
Montreal Cognitive Assessment | Assessments will be performed before the treatments, at 4 weeks after treatments, and at 8 weeks after treatments.
  Total score of this scale is 30 points, and patients with a score of ≥ 26 points are defined as normal.
Barthel Index | Assessments will be performed before the treatments, at 4 weeks after treatments, and at 8 weeks after treatments.
  The functional impairment is divided into mild (> 60 points), moderate (40-60 points), and severe level (≤ 40 points).

IPD SHARING:
Plan to Share IPD: No